CLINICAL TRIAL: NCT03237364
Title: Evaluation of Regional Lung Function in U.S. Soldiers With Suspected Iraq-Afghanistan War Lung Injury Using 19F MRI
Brief Title: Iraq- Afghanistan War Lung Injury Using 19F MRI (DIAL1001006)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Assistant Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00076112
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Constrictive Bronchiolitis; Iraq-Afganistan War Lung Injury Syndrome
Keywords: deployed in Iraq and/or Afghanistan
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Perfluorinated Gas/Oxygen Mixture — 19-Fluorine (19F) MRI of the lungs with 21%/79% Oxygen/Perfluorinated Gas, ≤ 25 liters, gas, single visit, < 1 hour
  Other Names: Perfluorinated Propane Imaging

SUMMARY:
The goal of this study is to evaluate the utilization of conventional 'thermally' polarized perfluorinated gases mixed with oxygen as an exogenous inert contrast agent to image the airway spaces in subjects with suspected lung disease, post deployment in Iraq and Afghanistan. This is an open label proof of concept study expanding on work here at Duke.

DETAILED DESCRIPTION:
There has been mounting evidence of respiratory problems related to military service in the Middle East especially in the past two decades. An overview by Flavo et al. summarizes studies not only of soldiers but evaluation of particulates from the Middle East in a number of animal models. While there have been some 'prospective' studies based on use of a standard evaluation protocol post deployment, the primary imaging modalities have been chest radiograph (most read as normal) and chest high resolution computed tomography (HRCT), neither of which have significant functional information. Standard pulmonary function testing (e.g. spirometry, lung volumes, diffusing capacity, bronchoalveolar lavage, as well as oscillatory resistance) were used in the STAMPEDE study, but only provide global functional information. The case study by King et al. included lung biopsy in a sub-cohort (n = 49) of soldiers with varying degrees of inhalation exposure during deployment. All biopsy samples were abnormal and some were consistent with constrictive bronchiolitis. Constrictive bronchiolitis is a non-reversible bronchiolar airway disease that is characterized by fibrosis of the bronchioles and can be challenging to diagnose without biopsy (it is also known by the term 'bronchiolitis obliterans'). The chest radiographs were normal in these subjects although about 25% of chest CT showed 'air trapping' or 'centrilobular nodules'. Pulmonary function testing in 39 soldiers with HRCT showed normal to near normal results in 32 of the subjects, with seven showing low diffusion capacity, obstruction and/or restriction. Clearly, neither global measures of lung function nor high resolution anatomic imaging are sensitive enough to avoid a biopsy to confirm diagnosis of constrictive bronchiolitis. We hypothesize that measures of regional lung function should provide additional information to aid in the diagnosis of WLI and may assist in the management of more difficult or advanced cases of WLI.

This is an open label study in up to 10 subjects being evaluated for post war lung injury. Each subject will receive up to 25 liters of inert perfluoropropane/oxygen gas mixtures as a contrast agent to visualize the airway and alveolar spaces in their lungs using 19F magnetic resonance imaging of inert gas/oxygen mixtures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial

  1. Outpatients of either gender, age > 18.
  2. Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed.)
  3. Women of childbearing potential must have a negative serum pregnancy test. This will be confirmed before participation in this investigational protocol.
  4. Subjects must have been deployed in Iraq and/or Afghanistan
  5. Subjects must have a strong clinical suspicion of a diagnosis of constrictive bronchiolitis based on clinical presentation and spirometry results

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the trial:

  1. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
  2. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
  3. Unable to receive gas mixture by breathing because of contraindications;
  4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Female; women at risk of pregnancy are required to have a confirmed negative urine pregnancy test at Screening if of childbearing potential prior to the MRI scan

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Lung Ventilatory Heterogeneity defined by parametric imaging with 19F perfluorinated gas/oxygen mixtures | one hour
  Fraction of lung with slow filling compartments compared to historic norms.

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University Medical Center, Department of Radiology
Locations (1):
- Duke Image Analysis Laboratory, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No